CLINICAL TRIAL: NCT01905410
Title: A Randomized, Double-blind, Single and Multiple Ascending Dose Escalation, Placebo-controlled Clinical Trial to Investigate Safety, Tolerability, and Pharmacokinetics of VVZ-149 Injection in Healthy Male Volunteers
Brief Title: Phase I Study to Investigate Safety, Tolerability, and Pharmacokinetics of VVZ-149 Injection
Acronym: P1_VVZ149IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-VVZ149-01
Record Dates: First submitted 2013-07-15; First posted 2013-07-23 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2013-07

CONDITIONS: Healthy
MeSH Terms: interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- single treatment - VVZ-149 Injection (Experimental): single ascending dose escalation
  * 0.25, 0.5, 1, 2, 4, 6, and 8 mg/kg Cohorts
  * 4 hours IV infusion
  Interventions: Drug: VVZ-149 Injection
- single treatment - placebo (Placebo Comparator): * The matching volume of placebo (water for injection) to each experimental cohort
  * 4 hours IV infusion
  Interventions: Drug: placebo
- multiple treatment - VVZ-149 Injection (Experimental): Based on the results of SAD trials, low and high dosage are determined for MAD trials.
  * high and low dosage
  * 4 hours IV infusion x 2 times/day x 3 days
  Interventions: Drug: VVZ-149 Injection
- multiple treatment - placebo (Placebo Comparator): * The matching volume of placebo (water for injection) to each experimental cohort
  * 4 hours IV infusion x 2 times/day x 3 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VVZ-149 Injection — VVZ-149 in water for injection
  Other Names: VVZ-149 Injection or Water for injection
  Arms: multiple treatment - VVZ-149 Injection; single treatment - VVZ-149 Injection
Drug: placebo — water for injection
  Other Names: VVZ-149 Injection or Water for injection
  Arms: multiple treatment - placebo; single treatment - placebo

SUMMARY:
VVZ-149 is a novel analgesic drug candidate that shows a potential analgesic activity inhibiting GlyT2 and 5HT2A simultaneously. There have been many efforts to develop single-target selective drugs to treat pain, but usually unsuccessful due to the lack of efficacy or limitations of single-target approach for new drug discovery. VVZ-149 is expected to have a dual-target activity, demonstrated having a synergism between GlyT2 and 5HT2A antagonistic activities to maximize an antinociceptive effect in the in vivo animal models. Now the investigators are developing VVZ-149 as an IV injection to treat post-operative pain.

The primary objective of this study is to evaluate a safety, tolerability and pharmacokinetic properties of VVZ-149 injection with placebo in healthy male volunteers. This Phase 1 study consists of a randomized, double-blind, placebo controlled, single and multiple ascending dose (SAD & MAD) escalation clinical trials.

DETAILED DESCRIPTION:
In this clinical study, the investigational drug product will be offered as an injectable form in a transparent glass vial that contains VVZ-149 dissolved by water for injection. When administered, the drug will be diluted by normal saline and will be given by intravenous infusion for 4 hours.

SAD study is planned that maximal 7 cohorts of healthy male subjects are administrated single dose of VVZ-149 injection or placebo. The planned groups for dose escalations were 0.25, 0.5, 1, 2, 4, 6, and 8 mg/kg groups. As a pilot study for safety in this first-in-human study, only 3 subjects received active drug are allocated to first two groups each, without subjects for placebo. For the following groups, 6 subjects for active drug and 2 for placebos are allocated after randomized.

MAD study is planned that 2 cohorts of 10 healthy male subjects each were administered multiple doses of VVZ-149 injection or placebo. The final doses of VVZ-149 injection will be determined later based on the results of SAD study. In each group, 7 subjects for active drug and 3 for placebos are allocated after randomized

ELIGIBILITY:
Subjects are eligible for the study if they met all the following Inclusion Criteria:

1. willingness to sign the written informed consent form (ICF)
2. 20~45 years, inclusive, healthy male
3. 50~90kg, inclusive, and within the 20% of ideal body weight
4. compatible at screening ( medical history, physical examination, vital signs, ECG, haematology, clinical chemistry, urinalysis)
5. sterility or keep an ascetic life or male subjects and their female sexual partners had to use a following contraception method during the study period *the medical contraception permissible method: condom, at least partner had to take the oral contraceptive over the 3 months or had to use the injection or insertion contraceptives, intrauterine device.

Subjects are to be excluded from participation if any of the following Exclusion Criteria:

1. Presence or history of diseases or abnormalities of liver, kidney, nervous system, respiratory system, endocrine system, or cardiovascular system. Presence or history of hemopathy or psychopathy (mood disorder, obsessive compulsive disorder etc.) Carrier of hepatitis virus in content of the liver disease, exclusive
2. History of hypersensitivity reactions significant clinically or hypersensitivity reaction to the investigational product, the drugs containing identical ingredient, or other drugs (aspirin, antibiotic etc.)
3. Family history of significant chronic pain disease or case of the immediate family (parent or brother) with chronic pain disease
4. Electrocardiogram QTc > 430 ms, PR interval > 200 msec, QRS interval > 120 msec, or any other clinically significant opinion at screening, exclusive
5. Any of following results in the Clinical laboratory at screening, exclusive

   * Exceed 1.25 times of the upper limit of the normal range of AST,AST
   * Exceed 1.5 times of the upper limit of the normal range of BUN, Cr
   * Out of normal range in Thyroid function (TSH, T4, FT4, T3) parameters
6. Abnormal blood pressure (systolic > 150 mmHg or < 90 mmHg, diastolic > 95 mmHg or < 60 mmHg) in vital signs at screening, exclusive
7. history of drug abuse, positive screen on the an alcohol breath test and an urine drug screening
8. Taking any ETC or oriental medicine within 2 weeks prior to drug administration, taking any OTC or vitamins within a week prior to drug administration, (but could participate in the study if other conditions are considered appropriate by the medical investigator)
9. Participation in a drug study (clinical trials) within 2 months prior to drug administration
10. Donation of whole blood within 2 months or blood component within a month or receiving a blood transfusion within a month prior to drug administration
11. Intake of more than 21 units per week (one unit of alcohol (10 g of pure alcohol) equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits), Unable to stop drinking during the study period
12. A smoker (if case of non-smoker to stop smoking within 3 months prior to drug administration, they could participate in this study) and positive screen on urine cotinine test.
13. Taking food and drink containing caffeine (coffee, tea, a carbonated drink, a coffee milk, and nutritious tonic etc) from 24 hours prior to hospitalization for clinical trial to discharge from hospital, Unable not to take them.
14. judged inappropriate because of medical, psychological, social and geographical conditions difficult to participate in the study or difficult to follow the treatment compliance or follow-up guidelines.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Adverse Events Appearance According to the NCI CTCAE V 4.02 | upto 8 days (SAD) / 13 days (MAD)
  According to the NCI CTCAE V 4.02, DLT (Dose Limiting Toxicity) is defined when it is applicable at least one criterion among following items
  * adverse event over CTCAE Grade 3
  * Any other significant toxicity according to the investigator's judgment
  Safety and Tolerability Measurements
  : physical examination, vital signs, 12-lead ECG, consecutive ECG and SpO2 monitoring, clinical laboratory tests(hematology, clinical chemistry, liver function, thyroid function, coagulation, urine analysis)

SECONDARY OUTCOMES:
Pharmacokinetic parameters | upto 2 days (SAD) / 5 days (MAD)
  Cmax, AUClast, AUCinf, Vd, MRT, t1/2, CL, fe, CLR

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Chung, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Sungnam-Si, Gyeonggi-do, South Korea